CLINICAL TRIAL: NCT02124850
Title: A Phase Ib Study of Neoadjuvant Immune Biomarker Modulation With Cetuximab Plus Motolimod and With Cetuximab Plus Motolimod Plus Nivolumab
Brief Title: A Phase Ib Study of Neoadjuvant of Cetuximab Plus Motolimod and Cetuximab Plus Motolimod Plus Nivolumab
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VRXP-A106
Record Dates: First submitted 2014-04-22; First posted 2014-04-28 (Estimated); Last update posted 2019-10-25 (Actual); Status verified 2019-10

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — VTX-2337; Cetuximab; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Motolimod plus cetuximab (Experimental): Cohort 1: motolimod plus cetuximab
  Interventions: Drug: Motolimod; Drug: Cetuximab
- Motolimod, cetuximab, and nivolumab (Experimental): Cohort 2: motolimod, cetuximab, and nivolumab
  Interventions: Drug: Motolimod; Drug: Cetuximab; Drug: Nivolumab

INTERVENTIONS:
Drug: Motolimod
  Other Names: VTX-2337
Drug: Cetuximab
  Other Names: Erbitux
Drug: Nivolumab
  Other Names: Opdivo
  Arms: Motolimod, cetuximab, and nivolumab

SUMMARY:
Protocol VRXP-A106 will enroll patients with Stage II-IVA head and neck cancer patients who will be treated with surgical resection. Cetuximab and motolimod (Cohort 1); and cetuximab, motolimod, and nivolumab (Cohort 2) will be administered for a 3-4 week period before surgery. The primary objective of the study is to determine the extent to which the administration of neoadjuvant motolimod plus cetuximab and motolimod plus cetuximab and nivolumab modulates immune biomarkers (NK, mDC and T cell activation as well as tumor infiltration and serum cytokines) in peripheral blood and head and neck cancer tumors. An exploratory objective of the study is to assess whether modulation of biomarkers as described above can predict anti-tumor response.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated stage II, III, or IVA histologically or cytologically confirmed squamous cell carcinoma of the head and neck
* Primary tumors of the oral cavity, oropharynx, hypopharynx, or larynx
* Macroscopic complete resection of the primary tumor must be planned
* Age ≥ 18 years
* ECOG performance status 0-1
* Adequate hematologic, renal and hepatic function
* Have signed written informed consent

Exclusion Criteria:

* Subjects who fail to meet inclusion criteria
* Primary tumors of the sinuses, paranasal sinuses, or nasopharynx, or unknown primary tumors
* Prior severe infusion reaction to a monoclonal antibody
* Pregnancy or breastfeeding
* Evidence of distant metastasis
* Any other malignancy active within 5 years except for non-melanoma skin cancer or carcinoma in situ of the cervix, DCIS or LCIS of the breast
* Prior history of head and neck cancer
* Prior therapy with motolimod, nivolumab, or other agents targeting PD-1/PD-L1
* Prior therapy targeting the EGFR pathway
* Acute hepatitis, known HIV, or active uncontrolled infection
* Patients with active autoimmune disease
* History of uncontrolled cardiac disease within prior 6 months
* Uncontrolled peptic or gastric ulcer disease, or gastrointestinal bleeding within prior 6 months
* Active alcohol abuse or other illness or circumstance that carries a likelihood of inability to comply with study treatment and follow-up or otherwise compromise the study's objectives
* Treatment with a non-approved or investigational drug within 30 days prior to Day 1 of study treatment
* Live vaccine within 30 days of planned start of study therapy
* History of pneumonitis or interstitial lung disease
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to nivolumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-10-28 (Actual); Primary Completion 2016-08-11 (Actual); Study Completion 2016-10-31 (Actual)

PRIMARY OUTCOMES:
The change in immune biomarkers including FcγR genotype, NK activation, tumor infiltration and serum cytokines, mDC, T cell activation, and tumor-antigen specific cytotoxic T lymphocyte induction. | change from baseline to up to 4 weeks

OTHER OUTCOMES:
Anti-tumor response | Change from baseline to pre-surgery

CONTACTS AND LOCATIONS:
Overall Officials: Amar Patel, MD, Study Director — Celgene
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Result] https://clincancerres.aacrjournals.org/content/clincanres/early/2017/11/28/1078-0432.CCR-17-0357.full.pdf